CLINICAL TRIAL: NCT05224063
Title: CRCNS US-France Research Proposal: Probing the Dorsolateral Prefrontal Cortex and Central Executive Network for Improving Neuromodulation in Depression
Brief Title: Probing the Dorsolateral Prefrontal Cortex and Central Executive Network for Improving Neuromodulation in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corey Keller, Associate Professor, Department of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 60980-2; R01MH129018 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Individualized CEN-targeted rTMS (Experimental): Individualized CEN-targeted rTMS will combine neuronavigated rTMS and single pulse TMS-EEG to identify the region of the dlPFC making the strongest connection with the parietal node of the CEN. First, regions of the dlPFC strongly connected to the parietal CEN will be identified by applying single TMS pulses in grid-like fashion to ROIs within the dlPFC. For each anatomical dlPFC subunit probed with TMS, the TMS-EEG response will be quantified in the parietal region of the CEN. The dlPFC subunit that demonstrates the strongest TMS-EEG response in parietal cortex will be chosen for rTMS. rTMS will last approximately 30 minutes (3000 pulses total) and will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS session for adverse events and/or side effects.
  Interventions: Device: Individualized CEN-targeted rTMS; Device: Sham rTMS
- Neuronavigated rTMS (Active Comparator): Neuronavigated rTMS will be delivered using neuro-navigation based on participants' own MRI images to target the dlPFC. rTMS will last approximately 30 minutes (3000 pulses total) and will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS session for adverse events and/or side effects.
  Interventions: Device: Neuronavigated rTMS; Device: Sham rTMS
- Scalp-targeted rTMS (Active Comparator): Scalp-targeted rTMS will be delivered using standard BEAM F3 targeting methodology to target the dlPFC. rTMS will last approximately 30 minutes (3000 pulses total) and will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the rTMS session for adverse events and/or side effects.
  Interventions: Device: Scalp-targeted rTMS; Device: Sham rTMS
- Sham rTMS (Sham Comparator): Sham rTMS will be delivered for one session to mimic active rTMS conditions. To maximize sham validity, both 1) a direction- sensor TMS coil will alert the operators to flip the coil if the wrong side is being used, and 2) low-intensity electrical stimulation to match the active rTMS frequency will be applied to scalp electrodes under the coil for sham and placed but not activated in the active arm. The rTMS coil will be positioned using neuro-navigation based on participants' own MRI images, mimicking active rTMS. Sham rTMS will last approximately 30 minutes (3000 pulses total) and will be delivered at 120% of the participant's motor threshold. Participants will be monitored during the sham rTMS session for adverse events and/or side effects.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Individualized CEN-targeted rTMS — Delivers patterned magnetic stimulation based on individualized CEN targeting
  Arms: Individualized CEN-targeted rTMS
Device: Neuronavigated rTMS — Delivers patterned magnetic stimulation based on MRI images
  Arms: Neuronavigated rTMS
Device: Scalp-targeted rTMS — Delivers patterned magnetic stimulation based on BEAM F3 targeting
  Arms: Scalp-targeted rTMS
Device: Sham rTMS — Delivers placebo magnetic stimulation

SUMMARY:
Depression is a highly prevalent condition characterized by persistent low mood, energy, and activity that can affect one's thoughts, mood, behavior, and sense of well-being. Repetitive transcranial magnetic stimulation (rTMS), a non-invasive neuromodulatory technique, is an effective treatment for depression when targeting the dorsolateral prefrontal cortex (dlPFC) of the central executive network (CEN). However, remission rates are suboptimal and individual methods to target the dlPFC are lacking. In this study, we will enroll 50 patients with major depression and in a single rTMS 'dose,' prospective, randomized, double-blind, cross-over design will assess whether rTMS targeted to an individual's central executive network (CEN) assessed by single pulse TMS can enhance network modulation. If successful, this work will lead to a clinical rTMS trial comparing this personalized targeting approach against standard rTMS.

DETAILED DESCRIPTION:
There is a critical need for more effective treatments for depression, which currently affect 20% of Americans during our lifetimes. Brain stimulation treatments, including repetitive transcranial magnetic stimulation (rTMS), represent the front line of innovative approaches by directly targeting and correcting specific dysfunctional brain networks. A core dysfunctional network in major depressive disorder is the fronto-parietal central executive network (CEN), a network critical for decision making and cognitive control. The CEN includes the dorsolateral prefrontal cortex (dlPFC), the target of FDA-cleared rTMS treatment for depression. rTMS to the dlPFC is thought to improve depression by modulating local dlPFC excitability and enhancing downstream CEN connectivity. However, our ability to probe the CEN and study this potential mechanism on an individual basis is critically lacking, likely contributing to suboptimal rTMS remission rates (20-40%). We hypothesize that the CEN connectivity is weakened in depression and can be maximally modulated by individualizing localization.

To test this hypothesis, in a single rTMS 'dose,' prospective, randomized, double-blind, cross-over design with 50 depressed patients, we will prospectively compare the strength, duration, and specificity of CEN modulation after a single session of dlPFC rTMS. These participants will be 18-65 years old and require a current major depressive disorder diagnosis assessed by Structured Clinical Interview for DSM5 (SCID-I62), with a PHQ9>10. Exclusion criteria includes contraindications for MRIs (e.g. implanted metal), history of head trauma with loss of consciousness, history of seizures, neurological or uncontrolled medical disease, active substance abuse, a history of suicide attempt in the past year, psychotic or bipolar disorders, a prior history of ECT or rTMS failure, and medications that substantially reduce seizure threshold (e.g., bupropion, clozapine).

Following the diagnostic session, participants will undergo a 30-minute MRI session to record structural brain data. For the following sessions, dlPFC will be targeted for each session using different methods and 10Hz dlPFC rTMS will be applied guided by (a) individualized CEN targeting, (b) structural MRI, (c) standard scalp targeting. For each condition, a single session of rTMS at standard parameters (10Hz, 5s on, 10s off, 3,000 total pulses, 15 min duration) will be performed and changes in CEN connectivity will be quantified using pre/post dlPFC-stimulated parietal TMS-evoked potentials (TEPs). The dlPFC will be targeted for rTMS using three methods: (a) MRI-guided with individual CEN optimization using TEPs, (b) MRI-guided alone, and (c) standard scalp targeting (Beam F3 method99). Additionally, a fourth session of sham rTMS will be applied to control for off-target effects. We hypothesize that while each active rTMS method (condition a-c) will suppress the p30 of the TEP in the CEN, optimized CEN localization using individual TEPs (condition a) will induce the strongest and most specific change in the CEN for the longest duration. Our primary outcome will be parietal p30 CEN modulation directly following rTMS. Secondary outcomes will assess parietal p30 changes in the parietal node of the CEN during rTMS (quantifying the p30 after the last pulse in each stimulation train) as well as 15 and 30 min following rTMS. We will also assess pre/post rTMS behavioral changes in attention with a standard continuous performance task and working memory using an N-back task, both of which have been implicated in the CEN and depression100,101. rTMS sessions will be triple-blinded to operator, participant, and statistician. rTMS sessions will be separated by at least two days to remove potential lasting effects >24 hours, and rTMS session order will be randomized and counterbalanced to reduce any potential bias.

Findings from this study will provide the basis for a clinical trial comparing rTMS treatment outcome using this personalized targeting approach against standard rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18 to 65
* Depression assessed through in-depth Structured Clinical Interview for DMS-5 (SCID-I)
* PHQ9 > 10 for disease severity
* Must comprehend English well to ensure adequate comprehension of the EEG and TMS instructions, and of clinical scales
* Right-handed
* No current or history of neurological disorders
* No seizure disorder or risk of seizures
* No use of PRN medication within 24 hours of the scheduled study appointment

Exclusion Criteria:

* Those with a contraindication for MRIs (e.g. implanted metal)
* Any unstable medical condition
* History of head trauma with loss of consciousness
* History of seizures
* Neurological or uncontrolled medical disease
* Active substance abuse
* Diagnosis of psychotic or bipolar disorder
* A prior history of ECT or rTMS failure
* Currently taking medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium)
* Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) / Electroencephalography (EEG) change | Up to 2 hours
  Change in TMS-EEG measures will be assessed before, during, and after each rTMS session. Specifically, the amplitude of the change 30ms after a single TMS pulse in the frontoparietal region will be quantified. Brain changes will be compared between CEN EEG-targeted, neuronavigated, scalp-targeted, and sham rTMS to identify the location, strength, and dose response of change for each condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States